CLINICAL TRIAL: NCT01744808
Title: A Phase 1 Study To Investigate the Pharmacokinetics of SR Formulations; and the Food Effect, Safety, Tolerance, Pharmacokinetic and Pharmacodynamic Profile Of 1 SR Formulation of EB-1020 In Young Healthy Subjects
Brief Title: A Study to Evaluate the Safety, Tolerance, and Pharmacokinetic and Pharmacodynamic Profile Of 1 SR Formulation of EB-1020
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurovance, Inc. (Industry)
Responsible Party: Sponsor
Organization: Euthymics BioScience, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: EB-1020-102
Record Dates: First submitted 2012-11-19; First posted 2012-12-07 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Normal, Healthy Volunteers
Keywords: Healthy; Normal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- EB-1020 SR1 (Active Comparator): Sustained release formulation
  Interventions: Drug: EB-1020 SR1
- EB-1020 SR2 (Active Comparator): Sustained Release Formulation
  Interventions: Drug: EB-1020 SR2
- EB-1020 SR3 (Active Comparator): Sustained Release Formulation
  Interventions: Drug: EB-1020 SR3
- EB-1020 IR (Active Comparator): Immediate Release Formulation
  Interventions: Drug: EB-1020 IR
- Placebo (Placebo Comparator): Placebo Formulation
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: EB-1020 IR — Immediate release
  Arms: EB-1020 IR
Drug: EB-1020 SR1 — sustained release
  Arms: EB-1020 SR1
Drug: EB-1020 SR2 — Sustained release
  Arms: EB-1020 SR2
Drug: EB-1020 SR3 — Sustained release
  Arms: EB-1020 SR3
Other: Placebo — Placebo formulation
  Arms: Placebo

SUMMARY:
To investigate whether there is a food-effect with oral administration with EB-1020 as well as to obtain information on the safety, and tolerability of EB-1020 in a range of doses.

DETAILED DESCRIPTION:
* To investigate the safety and tolerance of single doses of EB-1020 immediate release (IR) versus three sustained release (SR) formulations.
* To investigate the safety and tolerance of a single oral dose of a SR formulation of EB-1020 in the fed and fasted state.
* To investigate the safety, tolerance, and cognitive effects of multiple oral rising doses of a SR formulation of EB-1020.

Secondary Objectives

* To characterize the single dose and steady state pharmacokinetic profiles of EB-1020 SR formulations.
* To investigate the effect of food on the pharmacokinetic profile of EB-1020 SR following single oral doses.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-45 years inclusive
2. Body weight with the normal range for height (body mass index [BMI] between 19-30 kg/m2 inclusive)
3. If female, be of non-child bearing potential (surgically sterile, post-menopausal for 12 months or receiving a stable dose of implanted or injectable contraceptive for at least 3 months with last dose of injectable contraceptive within 2 months). Non-surgical menopause history must be confirmed by follicle-stimulating hormone (FSH) and luteinizing hormone (LH) levels as defined by established lab ranges.
4. Be in general good health without clinically significant medical history
5. Have clinical laboratory test results that are within the laboratory reference range; or if out of range are not clinically relevant and are acceptable to the Investigator and Sponsor medical representative
6. Negative Human Immunodeficiency Virus (HIV), Hepatitis B and Hepatitis Screening test
7. Able and willing to give written informed consent

Exclusion Criteria:

1. Receipt of any investigational agent or drug within 3 months of entry into the study
2. Use of prescription drugs within 4 weeks prior to first dosing. Subjects who have used over the counter medication excluding paracetamol, topical over the counter medications and routine vitamins but including megadose (intake of 20 to 600 times the recommended daily dose) vitamin therapy within 7 days of first dosing, unless agreed as non-clinically relevant by the Principal Investigator and Sponsor
3. A history of, or current evidence for, suicidal ideation, based upon clinical interview and a psychiatric questionnaire
4. A history of known or suspected seizures, spasms, infantile spasms, febrile convulsions, unexplained significant and recent loss of consciousness or history of significant head trauma with loss of consciousness or a family history (first degree relative) of epilepsy or seizures (fits)
5. A history of sleep problems in the last 3 months
6. A history of relevant atopy or drug hypersensitivity
7. A history (within the last 5 years) or evidence of alcohol or drug abuse. Subject who consume more than 14 units (female) or 21 (male) units of alcohol a week (unit = 1 glass (125 mL) of wine = 1 measure of spirits = ½ pint of beer) will also be ineligible
8. A positive urine test for drugs of abuse or alcohol at Screening or on the day of admittance to the Study Unit
9. A history of smoking in the last 3 months
10. Have a significant infection (such as influenza) or known inflammatory process on screening or admission
11. Have acute gastrointestinal symptoms at the time of screening or admission (e.g. nausea, vomiting, diarrhea, heartburn )
12. Have previously received EB-1020
13. Be vegetarians, vegans or have medical dietary restrictions
14. Any major surgical procedure within one month of entry into the study
15. Have difficulties communicating reliably with the Investigator or appear unlikely to co-operate with the requirements of the study in the investigator's judgment.
16. Any other condition which in the view of the Investigator is likely to interfere with study or put the subject at risk.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Cmax | up to 6 months
  Pharmacokinetic parameters
Tmax | up to 6 months
  Pharmacokinetic parameter
AUC | up to 6 months
  Pharmacokinetic parameter

SECONDARY OUTCOMES:
Effect of food on Cmax | up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Ltd., Melbourne, Victoria, Australia